CLINICAL TRIAL: NCT04382703
Title: Randomised Controlled Trial of a Self-Affirmation Theory-Based Intervention to Promote Hearing Aid Use
Brief Title: A Self-Affirmation Intervention to Promote Hearing Aid Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Kerry Ware, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 274086; IS-BRC-1215-20007 (Other Grant/Funding Number: NIHR Manchester Biomedical Research Centre)
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-05

CONDITIONS: Hearing Loss, Functional
MeSH Terms: conditions — Hearing Loss, Functional

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an intervention which is a questionnaire based with a self-affirmation embedded at the end of the questionnaire or they are assigned to a control group who undertake the same questionnaire minus the self-affirmation exercise.
Who Masked: Participant, Investigator
Masking Description: All postal questionnaires will be placed in opaque envelope and each envelope will be given a unique number, these unique numbers will be fed into a computerized list generator (www.random.org). The generated list will be used to put the questionnaires in batches for the audiologist to give to thier participants. The online version will automatically randomly assign participants to either the intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Given the associated questionnaire which has the embedded self-affirmation exercise.
  Interventions: Behavioral: Self-Affirmation Exercise
- Control (Active Comparator): Given the associated questionnaire without the embedded self-affirmation exercise.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Self-Affirmation Exercise — The self affirming exercise is as follow:
  The beginning to a sentence appears below. Below it are 4 different ways of completing the sentence. On the lines provided, please write out the beginning of the sentence and then complete it with 1 of the 4 options we have given you.
  If I feel threatened or anxious, then I will …………………………………..
  Options are as follows:
  think about the things I value about myself, remember things that I have succeeded in, think about what I stand for or think about things that are important to me
  Arms: Intervention
Behavioral: Control — Given a questionnaire minus the self affirming exercise
  Arms: Control

SUMMARY:
Hearing aids are the number one treatment for hearing loss and it is estimated that out of the 2 million of UK individuals who are supplied with hearing aids 1.4 million will use their hearing aids to varying degrees and the other 0.6 million will stop using their hearing aids altogether.

The proposed research is looking to improve hearing aid usage by using a self-affirmation intervention which lowers the threat of participants' ageing anxiety. The target of lowering participants' ageing anxiety to improve hearing aid use is because there is a stigma of hearing aids making people seem old and this stigma can make individuals resistant to wearing their hearing aids as they do not want to be seen in this light.

The current proposed research is an extension of a pilot study that was conducted in 2016 which found that a self-affirmation intervention may be useful in improving individuals' hearing aid usage. They randomly allocated 50 first-time hearing aid users either to a group that undertook a self-affirming exercise (e.g., "If I feel threatened or anxious, then I will think about the things I value about myself") or to a no-intervention control group. Consistent with the idea that self-affirmation helps people deal with threat, first-time hearing aid users reported significantly lower anxieties about ageing after self-affirming. Moreover, according to the data usage downloaded from their hearing aids (data-logging), the self-affirming group were found to have worn their hearing aids an average of two hours per day longer than the control group. Due to the limited number of participants, the effects of the intervention were not statistically significant. Nevertheless, the low cost and high potential public health "reach" alongside the effect size of d = 0.43 indicates that the intervention shows promise.

The main aim of this research is to re-test the self-affirmation intervention from the previous pilot study with a sufficiently large enough sample to answer the following "Does a self-affirmation intervention improve participant's hearing aid usage when compared to participants in the control group?

DETAILED DESCRIPTION:
Participants will be recruited through two NHS audiology clinics where they will be invited to participant in this study via an invitation letter either enclosed within their appointment letter or given to them at their audiology appointment. The information used to identify potential participants is that of their diagnoses (must be using or being supplied with hearing aids) . The audiology clinic staff will be identifying potential clients therefore it is believed that there is unlikely to be a breach of confidentiality. All participants will be sent a £10 shop-for-all voucher for participating in the second stage of the study (10-week post appointment) this will be sent to participants home after 6 months and this will include an invitation to a follow up questionnaire.

All prospective participants will be required to give written consent before being assigned to the study and those unable to do this will not be included. After consent is given participants will be allocated to either the intervention group or the control group. Procedure of the proposed study is as follows:

1. Each participant will be randomly assigned to either the control group or the intervention group. Blinding of both the participant and the researcher with regards to which group the participant has been assigned to will be achieved by all questionnaires being placed in opaque envelopes which will have a number printed on the front of the envelope. The numbers from the envelope will be placed in a computerised list generator and an order list of how they are to be administered will be produced. Alternatively participants can go online and the platform will randomly assign them to either the intervention or the control questionnaire.
2. Participants in both groups fill in a questionnaire which contain the following Scales: The Anxiety toward Ageing Scale (AAS), The Attitudes Toward Loss of Hearing Questionnaire (ATLH) and The Glasgow Benefit Hearing Aid Scale (GBHA) as well as a self-report question on their daily hearing aid use. The intervention group also undertake a self-affirmation exercise which is placed at the end of the questionnaire. This is expected to take 20-30 minutes.
3. Participants return 10 weeks later (post) and have their hearing aid usage downloaded (hours per day the aids were worn) from their hearing aids by an audiologist before subsequently filling in another questionnaire which again contains the AAS, ATLH, GBHA and a self- report question on their daily hearing aid use. This is expected to take 30-40 minutes.

3A: If it is not possible for the participant to come back for a follow up appointment the second questionnaire will be sent out postal to the participants address or an email with a hyperlink to the follow up questionnaire online will be sent to participants who previously completed the first questionnaire online.

4: Six months later participants are contacted via email ( hyperlink) or post to fill in an optional questionnaire containing the AAS, ATLH, GBHA and a self-report question on their daily hearing aid use which they send back to the researcher. This should take 20-30 minutes. If participants receive the follow up questionnaire through the post the shopping voucher will also be enclosed. Online participants will also receive their shopping voucher through the post.

5: A debrief form will be sent out via e-mail or post by the principal researcher 3 weeks after the follow up questionnaire was returned or alternatively if they decide to not to complete the follow up questionnaire the debrief will be sent 4 weeks after the initial questionnaire request was sent.

A G-power analysis was conducted to detect a small-moderate effect size (Cohen's D of 0.35) with 80% power at the 5% significance level which indicated that a sample of 260 participants (130 per group) would be required. This study will attempt to recruit 400 based on a similar pilot study having a 34% attrition rate. The data collection phase will continue until 260 participants have completed the 10 week follow up.

The study design is a mixed Design: Between-participants factor is condition (control vs intervention). Within-participants factor is time (pre-intervention vs post intervention (10-week) vs exit (6 month after post ). We will use a series of 2 (Intervention, control) x 3 ( pre-intervention, post intervention and exit) repeated ANOVA to assess to assess the outcome measures. If a small-moderate effect size (Cohen's d = 0.35) is found on any of the principle and secondary measures, then the Hayes PROCESS macro will be used to examine the possible mediating effects of the intervention on participants' hearing aid usage. If data is missing at the 10-week follow up the participant concerned will be excluded from the analysis at this point. The present study also has a longitudinal element and attrition at 6 months is expected. Any missing data will be addressed by using the "last observation carried forward technique".

All data such as contact details and ethnicity will be pseudonymised and kept in a separate, password protected file, in a restricted access folder on a secure University server. All paper copies of contact details and questionnaire data will be secured in Manchester University in a locked filing cabinet. Only the study team and regulatory monitoring and auditing authorities from the University of Manchester will have access to this data.

All the questionnaire data will be anonymised and kept in a separate, password protected file, in a restricted access folder on a secure University server. Only the study team and regulatory monitoring and auditing authorities from the University of Manchester will have access to this data.

The physical personal data copies will be kept until completion of the study then will be destroyed in accordance with University of Manchester regulations. All consent forms and questionnaire data are deemed as essential and this will be kept for 5 years to comply with University of Manchester regulations.

The current study will go through ethics approval with the National Health Service, Health Research Authority in the UK before it will be allowed to proceed. The study has already been through a preliminary ethics review at the University of Manchester.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+ receiving hearing aids for the 1st time already have hearing aids fitted able to provide written consent and can complete the simple questionnaire

Exclusion Criteria:

* Anyone younger than 18 anyone who does not wear a hearing aid anyone lacking in capacity to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-05 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-09-26 (Estimated)

PRIMARY OUTCOMES:
Hearing aid usage data from participants hearing aids | At the 10 weeks after baseline is taken
  The daily use of participants hearing aid use is pulled from their hearing aids data logging

SECONDARY OUTCOMES:
Participants self-reported measure of hearing aid use. | Baseline pre-intervention: 10 weeks after baseline: 34 weeks after baseline.
  Measured by asking participants "Thinking about how much you used your present hearing aid(s) over the past two weeks. On an average day, how many hours did you think you used the hearing aid(s)?"
Participants Anxiety toward Aging | Baseline pre-intervention: 10 weeks after baseline: 34 weeks after baseline.
  Will be measured by using The Anxiety Towards Ageing Scale (AAS; Lasher & faulkender,1993) this is a 20-question questionnaire. An example of the questions included is: "I expect to feel good about life when I am old" it is measured on a 7-point Likert scale 1= strongly disagree to 7= strongly agree.
Participants hearing loss/aid stigma. | Baseline pre-intervention: 10 weeks after baseline: 34 weeks after baseline.
  Will be measure using the subscale of "negative associations" from The Attitudes towards Loss of Hearing Questionnaire (Saunders & Cienkowski, 1996) there are 4 questions within this subscale an example is: "The thought of wearing a hearing aid makes me feel older." It is measured on a 7-point Likert scale 1= strongly disagree to 7= strongly agree.
Participants perceived benefit / satisfaction participants have for their hearing aids | Baseline pre-intervention: 10 weeks after baseline: 34 weeks after baseline.
  Will be measured by using the 4 standard questions presented on The Glasgow Benefit Hearing Aid scale (Gatehouse & Browning,1996). An example of these questions is "Please think about listening to the television with other family members or friends when the volume is adjusted to suit other people. Over the past two weeks, how much difficulty do you have in this situation?" It is answered on a 6-Likert scale 1= not applicable 2= Not at all and 6= Very much indeed.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Ware, Principal Investigator — The University of Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage CJ, Lees D, Lewis K, Munro KJ. Preliminary support for a brief psychological intervention to improve first-time hearing aid use among adults. Br J Health Psychol. 2017 Nov;22(4):686-700. doi: 10.1111/bjhp.12244. Epub 2017 May 9. PMID 28485483
- [Background] Overall, J. E., Tonidandel, S., & Starbuck, R. R. (2009). Last-observation-carried-forward (LOCF) and tests for difference in mean rates of change in controlled repeated measurements designs with dropouts. Social Science Research, 38(2), 492-503.